CLINICAL TRIAL: NCT00119210
Title: Bupropion for Smoking Cessation in Postpartum Women
Brief Title: Pilot Study of Bupropion for Smoking Cessation in Postpartum Non-breastfeeding Women
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: We were unable to recruit sufficient numbers of patients and decided that the study protocol was not feasible to implement
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Nancy Rigotti, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2004-P-001769; Grant #051794
Record Dates: First submitted 2005-07-05; First posted 2005-07-13 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2011-04

CONDITIONS: Tobacco Use Disorder
Keywords: Tobacco use cessation; Bupropion; Zyban; Puerperium
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use Cessation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): Sugar pill
  Interventions: Other: placebo
- Bupropion SR (Experimental)
  Interventions: Drug: Bupropion SR

INTERVENTIONS:
Drug: Bupropion SR
  Arms: Bupropion SR
Other: placebo
  Arms: Placebo

SUMMARY:
The purpose of this small preliminary study is to determine whether it is feasible to recruit women smokers who have just delivered a baby and are not breastfeeding into a study that would test whether starting bupropion, a smoking cessation medication, after a baby's birth helps a postpartum woman to stop smoking.

DETAILED DESCRIPTION:
Purpose: A pilot randomized double-blind placebo-controlled trial is testing the feasibility of conducting a full-scale trial of the efficacy of bupropion SR vs. placebo in non-breastfeeding postpartum women who smoked >1 cigarette in the last month of pregnancy and want to stop smoking. The study will estimate achievable enrollment and retention rates; estimate the effect size of the drug on tobacco abstinence; assess the tolerability of bupropion in postpartum women; and allow refinement of recruitment, retention, intervention, and assessment protocols.

Research Design: Pilot double-blind placebo-controlled randomized clinical trial.

Study Population: 40 postpartum women aged 18 years or older who smoked > 1 cigarette in the last month of pregnancy, want to stop smoking, and are not breastfeeding. Subjects will be recruited postpartum while hospitalized after delivery.

Intervention: Bupropion SR (or matching placebo) for 8 weeks, starting immediately post-delivery. The dose is 150 mg qd for one week then 150 mg bid for 7 weeks. All subjects will receive behavioral counseling delivered face-to-face during the post-delivery hospitalization and by telephone 4 times over 8 weeks.

Outcome Measures: (assessed at 2, 4, 8, and 12 weeks postpartum):

1. Study eligibility, recruitment, and retention rates (primary outcome).
2. Tobacco abstinence (7-day point prevalence nonsmoking by self-report and confirmed by saliva cotinine at 2 weeks, 8 weeks (end of drug treatment), and 12 weeks postpartum.
3. Postpartum weight loss and symptoms of depression and anxiety.
4. Tolerability of postpartum bupropion, assessed by medication adherence and adverse effects.

ELIGIBILITY:
Inclusion Criteria:

Postpartum women who:

* Smoked >1 cigarette in last month of pregnancy
* Deliver a baby at Brigham and Women's Hospital in Boston, MA
* Do not breastfeed or plan to breastfeed.
* Want to attempt to stop smoking

Exclusion Criteria:

* Age <18 years;
* Current use of bupropion or antidepressant;
* Current major depression or other severe psychiatric illness (e.g., schizophrenia, mania);
* Contraindication to use of bupropion;
* Illegal substance use in past 6 months;
* >1 drink/day of alcohol during pregnancy;
* Newborn with major congenital anomaly or <25 weeks' gestation;
* Inability to speak or read English;
* No telephone.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-03; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Proportion of women who are eligible for the study
Proportion of eligible women who enroll in the study
Proportion of enrolled women who complete the study

SECONDARY OUTCOMES:
Cotinine-verified 7-day tobacco abstinence at 2 weeks
Cotinine-verified 7-day tobacco abstinence at 8 weeks
Cotinine-verified 7-day tobacco abstinence at 12 weeks
Symptoms of depression at 2, 8, and 12 weeks postpartum
Symptoms of anxiety at 2, 8, and 12 weeks postpartum
Adherence to study drug at 2 and 8 weeks postpartum
Rate of adverse effects at 2 and 8 weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Rigotti, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States